CLINICAL TRIAL: NCT01331018
Title: Gene Transfer for Patients With Fanconi Anemia Complementation Group A (FANCA)
Brief Title: Gene Therapy for Fanconi Anemia
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Study ended early due to end of funding.
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Rocket Pharma Limited (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2097.00; NCI-2011-00202 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); RG9212015 (Other: Fred Hutch/University of Washington Cancer Consortium)
Record Dates: First submitted 2011-03-16; First posted 2011-04-07 (Estimated); Last update posted 2024-05-17 (Actual); Status verified 2024-05

CONDITIONS: Fanconi Anemia
MeSH Terms: conditions — Fanconi Anemia | interventions — Filgrastim; Granulocyte Colony-Stimulating Factor; Leukapheresis; Methylprednisolone; exifone; Medrol Veriderm; plerixafor; ferric pyrophosphate; Prednisone; deltacortene; prednylidene

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (hematopoietic stem progenitor cells) (Experimental): STEM CELL MOBILIZATION FOR CELL COLLECTION: Patients receive filgrastim SC BID for up to 6 days (on days 1-6 of mobilization). Patients receive plerixafor SC QD on days 4-6 of mobilization. PBSC count will be checked daily starting on day 4 of mobilization. Patients who have a PBSC count of >= 5 CD34+ cells/mcL will undergo up to 2 apheresis collections on consecutive days.
  BONE MARROW HARVEST FOR CELL COLLECTION: Patients with inadequate PBSC counts undergo bone marrow harvest for collection of stem/progenitor cells.
  REINFUSION: Patients receive methylprednisolone IV or prednisone PO on days -1 to 7 followed by a rapid taper over approximately 1 week and undergo reinfusion of genetically modified hematopoietic stem/progenitor cells on day 0.
  Interventions: Procedure: Bone Marrow Aspiration; Biological: Filgrastim; Biological: Genetically Engineered Hematopoietic Stem Progenitor Cells; Other: Laboratory Biomarker Analysis; Procedure: Leukapheresis; Drug: Methylprednisolone; Drug: Plerixafor; Drug: Prednisone

INTERVENTIONS:
Procedure: Bone Marrow Aspiration — Undergo bone marrow harvest
Biological: Filgrastim — Given SC
  Other Names: FILGRASTIM, LICENSE HOLDER UNSPECIFIED; G-CSF; Neupogen; r-metHuG-CSF; Recombinant Methionyl Human Granulocyte Colony Stimulating Factor; rG-CSF; Tevagrastim
Biological: Genetically Engineered Hematopoietic Stem Progenitor Cells — Undergo infusion of genetically modified hematopoietic progenitor cell therapy
  Other Names: Genetically Engineered HSPCs
Other: Laboratory Biomarker Analysis — Correlative studies
Procedure: Leukapheresis — Undergo leukapheresis
  Other Names: Leukocytopheresis; Therapeutic Leukopheresis
Drug: Methylprednisolone — Given IV
  Other Names: Adlone; Caberdelta M; DepMedalone; Depo Moderin; Depo-Nisolone; Duralone; Emmetipi; Esametone; Firmacort; Medlone 21; Medrate; Medrol; Medrol Veriderm; Medrone; Mega-Star; Meprolone; Methylprednisolonum; Metilbetasone Solubile; Metrocort; Metypresol; Metysolon; Predni-M-Tablinen; Prednilen; Radilem; Sieropresol; Solpredone; Summicort; Urbason; Veriderm Medrol; Wyacort
Drug: Plerixafor — Given SC
  Other Names: AMD 3100; JM-3100; Mozobil; SDZ SID 791
Drug: Prednisone — Given PO
  Other Names: .delta.1-Cortisone; 1, 2-Dehydrocortisone; Adasone; Cortancyl; Dacortin; DeCortin; Decortisyl; Decorton; Delta 1-Cortisone; Delta-Dome; Deltacortene; Deltacortisone; Deltadehydrocortisone; Deltasone; Deltison; Deltra; Econosone; Lisacort; Meprosona-F; Metacortandracin; Meticorten; Ofisolona; Orasone; Panafcort; Panasol-S; Paracort; PRED; Predicor; Predicorten; Prednicen-M; Prednicort; Prednidib; Prednilonga; Predniment; Prednisonum; Prednitone; Promifen; Servisone; SK-Prednisone

SUMMARY:
This clinical trial will access the toxicity and efficacy of infusion of gene modified cells for patients with Fanconi anemia (FA). Infusion of autologous patient blood stem cells that have been corrected in the laboratory by introduction of the normal gene may improve blood counts in patients with FA.

DETAILED DESCRIPTION:
OUTLINE:

STEM CELL MOBILIZATION FOR CELL COLLECTION: Patients receive filgrastim subcutaneously (SC) twice daily (BID) for up to 6 days (on days 1-6 of mobilization). Patients receive plerixafor SC once daily (QD) on days 4-6 of mobilization. Peripheral blood stem cell (PBSC) count will be checked daily starting on day 4 of mobilization. Patients who have a PBSC count of >= 5 CD34+ cells/mcL will undergo up to 2 apheresis collections on consecutive days.

BONE MARROW HARVEST FOR CELL COLLECTION: Patients with inadequate PBSC counts undergo bone marrow harvest for collection of stem/progenitor cells.

REINFUSION: Patients receive methylprednisolone intravenously (IV) or prednisone orally (PO) on days -1 to 7 followed by a rapid taper over approximately 1 week and undergo reinfusion of genetically modified hematopoietic stem/progenitor cells on day 0.

After completion of study treatment, patients are followed up periodically for 15 years.

ELIGIBILITY:
Inclusion Criteria:

* FA demonstrated by a positive test for increased sensitivity to chromosomal breakage with mitomycin C or diepoxybutane performed by a Clinical Laboratory Improvement Amendments (CLIA) or College of American Pathologists (CAP) approved laboratory
* FA complementation group A as determined by somatic cell hybrids, molecular characterization, western blot analysis, acquisition of mitomycin C resistance after in vitro lentiviral transduction with a vector bearing the complementary deoxyribonucleic acid (cDNA) for Fanconi complementation group A, or other clinically certified method of complementation group analysis
* Bone marrow analysis demonstrating normal cytogenetics, and no more than 5% of cells with a single clonal abnormality by fluorescence in situ hybridization (FISH) for myelodysplastic syndrome (MDS) panel within 3 months of stem cell collection
* Signed informed consent by the patient or legally authorized representative
* Absolute neutrophil count >= 0.5 x 10^9/L
* Hemoglobin >= 8 g/dL
* Platelet count >= 20 x 10^9/L and able to achieve a platelet count of >= 50 x 10^9/L with transfusion support
* Adequate hepatic function with aspartate aminotransferase (AST) and alanine aminotransferase (ALT) < 5 x upper limit of normal (ULN)
* Adequate renal function with creatinine (Cre) =< 1.5; if greater, then glomerular filtration rate (GFR) > 60 mL/min/1.73 m^2 as calculated by the Modification of Diet in Renal Disease equation
* Adequate pulmonary function with corrected diffusion capacity of carbon monoxide (DLCO) > 50% in those for whom this study can be performed
* For subjects < 17 years of age, Modified Lansky Play-Performance Score of >= 70%; for subjects 17 and older, Karnofsky score of >= 70%

Exclusion Criteria:

* Non-hematopoietic malignancy where the expected survival is less than 2 years
* Myelodysplastic syndrome as defined by World Health Organization (WHO) criteria
* Acute myeloid leukemia as defined by WHO criteria
* Pregnancy or lactation; females of childbearing potential and males who are admitted to the study will be advised that the study procedures and study drugs may be teratogenic, and they will be required to take adequate measures to prevent conception for the duration of the study
* Concurrent enrollment in any other study using an investigational drug
* Physical or emotional status that would prevent informed consent, protocol compliance, or adequate follow-up
* Patients for whom an human leukocyte antigen (HLA) matched sibling donor bone marrow transplant is being actively pursued will not be eligible for study until it is determined that no sibling donor is available or that a stem cell transplant is not feasible during the time the patient might be on study

  * No patient will be included in this study as an alternative to a clinically indicated HLA matched sibling donor stem cell transplant
  * If an HLA matched sibling donor is identified, but stem cell or marrow collection is not feasible (e.g., donor is in utero, is a newborn from whom cord blood was not collected, or is unable to undergo a donation procedure because of ill health), a patient may be included in the study at the discretion of the investigators
* Significant associated diseases including documented human immunodeficiency virus (HIV) infection, uncontrolled hypertension (diastolic blood pressures > 95%ile for age), unstable angina, congestive heart failure (> New York [NY] class II), poorly controlled diabetes (hemoglobin A1c [Hgb A1c] > 7%), coronary angioplasty within 6 months, myocardial infarction within the last 6 months, or uncontrolled atrial or ventricular cardiac arrhythmia, abnormal coagulation, persistent abnormal urinalysis reflecting intrinsic renal disease
* Active ongoing viral, bacterial, or fungal infection

Min Age: 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2012-02-22 (Actual); Primary Completion 2024-02-15 (Actual); Study Completion 2024-02-15 (Actual)

PRIMARY OUTCOMES:
Toxicity of gene transfer | Up to 15 years
  Adverse events will be graded by Common Terminology Criteria for Adverse Events (CTCAE), version 4.
Hematological and non-hematological organ toxicity | Up to 15 years
  Adverse events will be graded by CTCAE, version 4.
Development of insertional mutagenesis or hematologic malignancy | Up to 15 years
  Adverse events will be graded by CTCAE, version 4.
Development of replication competent lentivirus | Up to 15 years
  Adverse events will be graded by CTCAE, version 4.

SECONDARY OUTCOMES:
Efficacy of G-CSF and plerixafor mobilization in Fanconi anemia (FA) patients | Up to 6 days
Efficacy of lineage depletion of bone marrow or mobilized cell product | Up to 15 years
Transduction efficiency | Day 0
  After completion of lentiviral transduction, the percent gene modified cells will be determined by molecular studies.
Detectable levels of transduced cells in blood and marrow | Up to 1 year
  Blood and bone marrow samples will be assayed by real-time quantitative polymerase chain reaction.
Improved blood counts | Up to 15 years
  Complete blood counts will be monitored, initially weekly, then monthly during the first year, then quarterly during the 2nd year after infusion.
Demonstrable functional expression by growth of recipient cells in mitomycin C | 3 months
  Blood and bone marrow cells will be assayed for viability of cultured cells and hematopoietic colonies in the presence of the chemotherapy drug and deoxyribonucleic acid crosslinking agent, mitomycin C.

CONTACTS AND LOCATIONS:
Overall Officials: Hans-Peter Kiem, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States